CLINICAL TRIAL: NCT04844736
Title: Pilot Study: Testing the Feasibility of a Simplified Workflow for Lung Cancer Radiation Target Review With Radiology
Brief Title: Testing the Feasibility of a Simplified Workflow for Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00072886; WFBCCC 01221 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2021-04-12; First posted 2021-04-14 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiology Treatment Planning/Review (Other): After patient consultation and enrollment, the patient will undergo routine CT simulation to initiate the radiation treatment planning process. The treating physician will contour the gross tumor volume (GTV) including the involved primary lung tumor and/or the involved lymph nodes. If the initial radiology review reflects concern for inadequate target volume delineation, the case will be flagged for multidisciplinary discussion between the radiation oncologist and radiologist.
  Interventions: Procedure: CT Simulation

INTERVENTIONS:
Procedure: CT Simulation — Patient will undergo routine CT simulation to initiate radiation treatment planning process. For the purposes of this study, the day of CT simulation "mapping scan" will be counted as day 0. After the patient completes the CT simulation scan, the CT images and plan/structure files will be sent to the treatment planning system. The treating physician will contour the gross tumor volume (GTV) including the involved primary lung tumor and/or the involved lymph nodes.

SUMMARY:
The purpose of this research study is to see if adding an "extra" check by formal radiology review is possible without disrupting the normal processes that take place to develop and prepare a safe radiation treatment plan for patients.

DETAILED DESCRIPTION:
Primary Objectives: The primary objective will be to demonstrate the feasibility of radiology completing real time review of radiation oncology treatment plans within 4 business days of the date of CT simulation (defined as day = 0). If 50% of plans can be reviewed by any member of the thoracic radiology team (Includes radiology PI and co-investigators) and feedback is submitted to radiation oncology with Appendix D within 4 business days of the date of simulation, then we will consider this workflow feasible.

Secondary Objectives:

* Our primary secondary objective will be to estimate the proportion of patients whose RT plans are changed as a result this workflow.
* For patients whose radiation therapy plans are changed as a result this workflow, determine the absolute and percentage volume changes in the gross tumor volume, clinical target volume and planning target volume as a result of these changes implemented.
* For patients whose radiation therapy plans are changed as a result of this workflow: determine if recommended changes in the gross tumor volume resulted in improved dosimetry to surrounding normal structures. Specifically, determine the absolute and percentage changes in the dose delivered to the lungs (V5, V10, V20) and esophagus (mean, V60) as a result of changes in the gross tumor volume.
* For patients whose radiation therapy plans are changed as a result of this workflow, determine if changes led to treatment delays from their standard planned start date.
* For patients whose radiation therapy plans are changed as a result of this workflow, to describe the most common types of changes recommended (i.e. modification of parenchymal lung volumes, missing involved lymph nodes, covering too much normal tissue in the gross tumor volume).
* Determine whether acute esophagitis incidence changed in our entire sample as a result of this review during treatment and within 4 weeks following treatment, compared to institutional historical control databases of patients treated without formal radiology review.
* Determine whether tumor response at 4 weeks post treatment differs in our entire sample compared to institutional historical control databases of patients treated without formal radiology review.

ELIGIBILITY:
Inclusion Criteria:

* Disease that is being treated as locally advanced non-small cell lung cancer (NSCLC) or limited stage small cell lung cancer (SCLC). Specifically, AJCC 8th edition staging with T3 or T4 and/or N1-3 disease. Patients with unclear pathology who are being treated clinically as non-small cell lung cancer or as limited stage small cell lung cancer are eligible.
* Plan for radiotherapy to be delivered with curative intent per the treating radiation oncologist in the Wake Forest Baptist Comprehensive Cancer Center Department of Radiation Oncology.

Exclusion Criteria: Not being treated with radiation, or being treated with non-curative intent per the treating radiation oncologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Number of Completed Radiation Treatment Plans Reviewed | Within four days after CT simulation
  Completed initial radiology review within 4 business days after the date of CT simulation will be calculated using summary statistics including count (frequency) using a 95% confidence interval.

SECONDARY OUTCOMES:
Number of Patients Whose Radiation Treatment Plans Changed | 4 days
  Will be calculated using summary statistics including count (frequency) and corresponding 95% confidence intervals.
Changes in Volumes After Radiation Treatment Changes - Gross Tumor Volume | 4 days
  For patients whose radiation therapy plans are changed, the change in volume (in centimeters cubed) of gross tumor volume (GVT) before and after the recommended change is made will be summarized using mean and standard deviation and median range.
Changes in Volumes After Radiation Treatment Changes - Clinical Tumor Volume | 4 days
  For patients whose radiation therapy plans are changed, the change in volume (in centimeters cubed) of clinical target volume (CTV) before and after the recommended change is made will be summarized using mean and standard deviation and median range.
Changes in Volumes After Radiation Treatment Changes - Planning Tumor Volume | 4 days
  For patients whose radiation therapy plans are changed, the change in volume (in centimeters cubed) of planning target volume (PTV) before and after the recommended change is made will be summarized using mean and standard deviation and median range.
Changes in Dose Delivered After Radiation Treatment Changes to the Lungs | 4 days
  For patients whose RT plans are changed, the change in the dose delivered to the lungs (V5, V10, V20) will be summarized using mean (standard deviation) and median (range).
Changes in Dose Delivered After Radiation Treatment Changes to the Esophagus | 4 days
  For patients whose RT plans are changed, the change in the dose delivered to the and esophagus (mean, V60) will be summarized using mean (standard deviation) and median (range).
Number of Patients Who's Treatment Starts are Delayed | 4 days
  For patients whose radiation therapy plans are changed: the proportion of treatment starts that are delayed from the initial planned start day due to the application of recommended changes will be calculated using summary statistics including count (frequency)
Number of Changes Recommended by the Radiation Therapy Quality Assurance Conference (RT QAC) | 4 days
  Will be calculated using summary statistics including count (frequency) and will also be captured in full qualitative form.
Number of Patients with Acute Esophagitis | 4 weeks after completion of therapy
  Will be reported using descriptive statistics (mean, median, standard deviations, proportions, and 95% confidence intervals) and will also be compared to the historical institutional control incidence and severity of esophagitis using 1-sample z-tests and 1-sample tests of proportions (considering historical control as "population parameter.")
Cancer Response | 1 month after completion of therapy
  Will be assessed by radiology on imaging and will be summarized using frequencies and proportions. Proportion of those with positive response will be compared to historical institution control using a 1-sample test of proportions (considering historical control as "population parameter.").

CONTACTS AND LOCATIONS:
Overall Officials: Michael Farris, MD, Principal Investigator — Wake Forest Baptist Comprehensive Cancer Center
Locations (4):
- United States (4):
  - High Point Medical Center, High Point, North Carolina
  - Wake Forest Baptist Health - Lexington, Lexington, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wake Forest Baptist Health Sciences, Winston-Salem, North Carolina

REFERENCES:
- [Derived] Farris MK, Razavian NB, Hughes RT, Ververs JD, Snavely AC, Leyrer CM, Tye KE, Allen LF, Pacholke HD, Weaver KE, Bunch PM, Chan MD, Clark H, Puthoff G, Farris JC, Steber CR, Wentworth S, Levine BJ, Nightingale CL, Ponnatapura J. Bridging the Communication Gaps: A Prospective Single-Arm Pilot Study Testing the Feasibility of Interdisciplinary Radiotherapy Planning in Locally Advanced Lung Cancer. Acad Radiol. 2023 Nov;30(11):2566-2573. doi: 10.1016/j.acra.2023.01.019. Epub 2023 Feb 8. PMID 36759296

DOCUMENTS (1):
  • Informed Consent Form (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT04844736/ICF_000.pdf